CLINICAL TRIAL: NCT04399239
Title: A Multicenter, Single Arm, Prospective, Open-Label, Staged Study of the Safety and Efficacy of the AuriNovo Construct for Auricular Reconstruction in Subjects With Unilateral Microtia
Brief Title: AuriNovo for Auricular Reconstruction
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company decision, not safety related.
Sponsor: 3DBio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3DBio12A2020
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2023-05

CONDITIONS: Microtia
Keywords: ear reconstruction
MeSH Terms: conditions — Congenital Microtia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- AuriNovo (Experimental): AuriNovo is a patient-specific, biologically natural, supportive base for surgical reconstruction of the external ear (auricle) in people born with microtia Grades II-IV. The construct is a 3D-bioprinted collagen hydrogel scaffold encapsulating the patient's own auricular cartilage cells (chondrocytes). The construct is printed in a size and shape that matches the contralateral ear for implantation into the patient.
  Interventions: Combination Product: AuriNovo

INTERVENTIONS:
Combination Product: AuriNovo — AuriNovo is a patient-specific, biologically natural, supportive base for surgical reconstruction of the external ear (auricle) in people born with microtia Grades II-IV. The construct is a 3D-bioprinted collagen hydrogel scaffold encapsulating the patient's own auricular cartilage cells (chondrocytes). The construct is printed in a size and shape that matches the contralateral ear for implantation into the patient.
  Other Names: AACC

SUMMARY:
AuriNovo provides a patient-specific, biological construct for use in the surgical reconstruction of the external ear in people born with microtia Grades II-IV. This Phase 1 / 2A study is being conducted to collect preliminary safety data on microtic ear reconstruction using AuriNovo, fine-tune technical, logistical, surgical, and post-surgical care aspects related to implantation, and to gather preliminary efficacy data including short- and longer-term in vivo duration and biological status of the implant.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric children 6-11, adolescents 12-16, or adults 17-25 years old
2. Born with unilateral microtia Grade II, III, or IV
3. No previous surgical procedure for auricular reconstruction
4. Have undergone an audiological assessment prior to enrollment and surgeon confirmation that study participation will not preclude future hearing correction options
5. Normal or near normal hairline position
6. Able to adhere to the follow-up schedule and post-surgery care instructions
7. Ability for the subject and/or guardian to understand and give informed consent
8. Healthy subjects with no history of cancer, problematic wound healing, or immune disorders

Exclusion Criteria:

1. Previous cochlear implant surgery
2. Patients with prior surgery in the temporal, parietal, or mastoid regions of the affected side that resulted in scarring that may affect the outcome of microtia reconstruction surgery.
3. Sensitivity to broad-spectrum aminoglycoside antibiotics containing any of the following: streptomycin, gentamycin tobramycin, amikacin, kanamycin, neomycin, or plazomicin.
4. Sensitivity to materials of porcine origin including pork products. For subjects with no known exposure to porcine materials including pork products, sensitivity as confirmed at baseline through a positive porcine skin sensitivity test.
5. Patients previously diagnosed/evaluated for any of the following syndromes:

   1. CHARGE (Coloboma, Heart defect, choanal Atresia, Retarded growth and development, Genital hypoplasia, Ear anomalies) syndrome,
   2. Branchio-oto-renal (BOR) syndrome
   3. Patients with renal dysfunction of any etiology
6. Patients with abnormal renal function determined at baseline with a blood test.
7. Patients with a history of keloid formation.
8. Patients with current skin infection.
9. Patients on immunosuppressants.
10. Any cognitive disorders where the patient would not be able to complete subject assessment questionnaires.
11. Lifestyle activities likely to affect healing or ability to adhere to the protocol (e.g., active contact sports and protective gear interferes with wearing post-operative ear protection)
12. Patients requiring chronic use of any headgear (e.g., CPAP) that would interfere with the ability to wear post-operative ear protection.
13. Pregnant females (a negative pregnancy test is required for females with reproductive potential)
14. Female patients who are nursing/lactating
15. Patients of reproductive potential (male and female) unwilling to use effective contraception during the first post-operative year.

    For this first-in-human study, microtia patients with significant craniofacial asymmetries or deformities from other syndromes will be excluded in order to aid initial assessments of efficacy of AuriNovo. The following syndromes or conditions are additional exclusion factors:
16. Treacher-Collins Syndrome
17. Nager Syndrome
18. Goldenhar syndrome or hemifacial microsomia plus an occlusal cant of 20 degrees or greater
19. Absence of vertical ramus (as diagnosed on physical exam or CT)
20. Absence of zygoma (as diagnosed on physical exam or CT)
21. Significant orbital asymmetry or micro-ophthalmia (as diagnosed on physical exam or CT)

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Safety through assessment of AEs | 3 months
  Safety data will be collected on AE type, frequency and severity, treatment, and the time to resolution.
Efficacy as measured through overall satisfaction scores | 3 months
  Data will be collected to determine the suitability of the AACC to support reconstruction of the outer ear in microtia patients. The following will be used to determine satisfaction;
  - Surgical Outcomes Questionnaire (scores range from 15 (lowest satisfaction) to 75 (highest satisfaction))
Efficacy as measured through overall satisfaction scores | 3 months
  Data will be collected to determine the suitability of the AACC to support reconstruction of the outer ear in microtia patients. The following will be used to determine satisfaction;
  - FACE-Q Kids Questionnaire (scores range from 74 (lowest satisfaction) to 296 (highest satisfaction))

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - John Reinisch, MD, Beverly Hills, California
  - Microtia-Congenital Ear Deformity Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No